CLINICAL TRIAL: NCT07229209
Title: Oral Contraceptive Pills Versus Levonorgestrel-Releasing Intrauterine System for the Management of Niche-Related Abnormal Uterine Bleeding: A Prospective Open-Label Randomized Controlled Trial
Brief Title: Oral Contraceptive Pills Versus Levonorgestrel-Releasing Intrauterine System for Niche-Related Abnormal Uterine Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Latif Ahmed Alnezamy, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC10-2-2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Abnormal Uterine Bleeding; Cesarean Section Complications; Uterine Scar
Keywords: cesarean scar defect; Uterine niche; abnormal uterine bleeding; oral contraceptive pills; levonorgestrel intrauterine system; randomized controlled trial
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Masking Description: Because of the nature of the interventions, blinding was not feasible; hence, the trial was open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined oral contraceptive pill group (Active Comparator): Participants received a monophasic combined oral contraceptive pill containing 0.03 mg ethinyl estradiol and 3 mg drospirenone (Technospiron® 0.03/3 mg, Technopharm, Egypt), taken for 21 days starting on day 2 of menstruation for six consecutive cycles.
  Interventions: Diagnostic Test: transvaginal ultrasonography; Drug: monophasic combined oral contraceptive pill
- levonorgestrel-releasing intrauterine system group (Active Comparator): Participants received a 52 mg levonorgestrel-releasing intrauterine system (Mirena®, Bayer, Oy Finland), inserted under transvaginal ultrasound guidance within the first three days of menstruation for 6 months.
  Interventions: Diagnostic Test: transvaginal ultrasonography; Device: 52 mg levonorgestrel-releasing intrauterine system

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasonography — At baseline and at 6 months after the start of treatment, transvaginal ultrasonography was performed to assess residual myometrial thickness, niche depth, length, and width.
Drug: monophasic combined oral contraceptive pill — Participants received a monophasic combined oral contraceptive pill containing 0.03 mg ethinyl estradiol and 3 mg drospirenone (Technospiron® 0.03/3 mg, Technopharm, Egypt), taken for 21 days starting on day 2 of menstruation for six consecutive cycles.
  Other Names: Technospiron
  Arms: combined oral contraceptive pill group
Device: 52 mg levonorgestrel-releasing intrauterine system — Participants received a 52 mg levonorgestrel-releasing intrauterine system (Mirena®, Bayer, Oy Finland), inserted under transvaginal ultrasound guidance within the first three days of menstruation for 6 months.
  Other Names: Mirena
  Arms: levonorgestrel-releasing intrauterine system group

SUMMARY:
The purpose of the study is to compare the clinical efficacy and niche morphological changes following treatment with combined oral contraceptive pills (OCPs) versus a levonorgestrel-releasing intrauterine system (LNG-IUS) in women with symptomatic uterine niche-related abnormal uterine bleeding (AUB).

DETAILED DESCRIPTION:
After eligibility and consenting, participants were randomized in a 1:1 ratio using a computer-generated block randomization list (block size of six). Allocation concealment was maintained using sequentially numbered, opaque, sealed envelopes, which were opened after consent.

All participants had a transvaginal ultrasound-confirmed uterine niche ≥2 mm in depth. Residual myometrial thickness, niche depth, length, and width were assessed.

* OCP group: Participants received a monophasic combined oral contraceptive pill containing 0.03 mg ethinyl estradiol and 3 mg drospirenone (Technospiron® 0.03/3 mg, Technopharm, Egypt), taken for 21 days starting on day 2 of menstruation for six consecutive cycles.
* LNG-IUS group: Participants received a 52 mg levonorgestrel-releasing intrauterine system (Mirena®, Bayer, Oy Finland), inserted under transvaginal ultrasound guidance within the first three days of menstruation for 6 months.

Both treatments were provided free of charge. Participants could switch to the alternative method upon study completion. Because of the nature of the interventions, blinding was not feasible; hence, the trial was open-label. Assessments were performed at baseline and at 1, 3, and 6 months. Participants recorded:

* Number of days of postmenstrual/intermenstrual spotting
* Total bleeding duration per cycle
* Pelvic pain and dysmenorrhea scores (10-point visual analogue scale)
* Sexual well-being (5-point Likert scale)
* Treatment satisfaction (satisfied/very satisfied vs. other responses)
* Adverse events, complications, and reasons for discontinuation (including LNG-IUS expulsion) At 6 months, transvaginal ultrasonography was repeated to assess residual myometrial thickness, niche depth, length, and width.

ELIGIBILITY:
Inclusion Criteria:

* women with at least one previous cesarean section.
* presenting with postmenstrual or intermenstrual bleeding for ≥3 consecutive cycles lasting ≥2 days, and a total bleeding duration >7 days per cycle.
* All participants had a transvaginal ultrasound-confirmed uterine niche ≥2 mm in depth.

Exclusion Criteria:

* pregnancy
* malignancy
* other identifiable causes of abnormal uterine bleeding
* abnormal cervical cytology
* cervicitis
* pelvic inflammatory disease
* endometrial polyps
* uterine fibroids
* contraindications to either combined oral contraceptive pill or levonorgestrel-releasing intrauterine system
* desire for pregnancy
* refusal to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Number of days of postmenstrual/intermenstrual spotting | at baseline and at 1, 3, and 6 months
  Participants recorded this on a paper Menstrual Diary charts

SECONDARY OUTCOMES:
Total bleeding duration per cycle | at baseline and at 1, 3, and 6 months
  Participants recorded this on a paper Menstrual Diary charts
Pelvic pain scores | at baseline and at 1, 3, and 6 months
  Participants recorded this on 10-point visual analogue scale where 0 means no pain and 10 means intense pain.
dysmenorrhea scores | at baseline and at 1, 3, and 6 months
  Participants recorded this on 10-point visual analogue scale where 0 means no pain and 10 means intense pain.
Sexual well-being | at baseline and at 1, 3, and 6 months
  Participants recorded this on 5-point Likert scale where 1 means never or not at all and 5 means always or extremely.
Treatment satisfaction | at 1, 3, and 6 months
  Participants recorded this as Yes if they are satisfied/very satisfied or No if they are neutral or dissatisfied
Adverse events | at 1, 3, and 6 months
  Participants reported this to the main investigator via telephone calls
complications | At 1, 3, and 6 months
  Participants reported this to the main investigator via telephone calls
reasons for discontinuation | At 1, 3, and 6 months
  Participants reported this to the main investigator via telephone calls

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ALNEZAMY, MD, Principal Investigator — Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Locations (1):
- Benha Univesity Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naji O, Abdallah Y, Bij De Vaate AJ, Smith A, Pexsters A, Stalder C, McIndoe A, Ghaem-Maghami S, Lees C, Brolmann HA, Huirne JA, Timmerman D, Bourne T. Standardized approach for imaging and measuring Cesarean section scars using ultrasonography. Ultrasound Obstet Gynecol. 2012 Mar;39(3):252-9. doi: 10.1002/uog.10077. PMID 21858885
- [Background] Tulandi T, Cohen A. Emerging Manifestations of Cesarean Scar Defect in Reproductive-aged Women. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):893-902. doi: 10.1016/j.jmig.2016.06.020. Epub 2016 Jul 5. PMID 27393285
- [Background] Vikhareva Osser O, Valentin L. Clinical importance of appearance of cesarean hysterotomy scar at transvaginal ultrasonography in nonpregnant women. Obstet Gynecol. 2011 Mar;117(3):525-532. doi: 10.1097/AOG.0b013e318209abf0. PMID 21343754
- [Background] Donnez O. Cesarean scar defects: management of an iatrogenic pathology whose prevalence has dramatically increased. Fertil Steril. 2020 Apr;113(4):704-716. doi: 10.1016/j.fertnstert.2020.01.037. PMID 32228874
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Result] Stavridis K, Balafoutas D, Vlahos N, Joukhadar R. Current surgical treatment of uterine isthmocele: an update of existing literature. Arch Gynecol Obstet. 2025 Jan;311(1):13-24. doi: 10.1007/s00404-024-07880-w. Epub 2024 Dec 16. PMID 39680143
- [Result] Klein Meuleman SJM, Min N, Hehenkamp WJK, Post Uiterweer ED, Huirne JAF, de Leeuw RA. The definition, diagnosis, and symptoms of the uterine niche - A systematic review. Best Pract Res Clin Obstet Gynaecol. 2023 Aug;90:102390. doi: 10.1016/j.bpobgyn.2023.102390. Epub 2023 Jul 15. PMID 37506497
- [Result] Murji A, Sanders AP, Monteiro I, Haiderbhai S, Matelski J, Walsh C, Abbott JA, Munro MG, Maheux-Lacroix S; International Federation of Gynecology and Obstetrics (FIGO) Committee on Menstrual Disorders and Related Health Impacts. Cesarean scar defects and abnormal uterine bleeding: a systematic review and meta-analysis. Fertil Steril. 2022 Oct;118(4):758-766. doi: 10.1016/j.fertnstert.2022.06.031. Epub 2022 Aug 17. PMID 35985862
- [Result] You SH. The symptomatic cesarean scar defect with oral contraceptive pills treatment following evacuation of a cesarean scar pregnancy. Taiwan J Obstet Gynecol. 2023 Jan;62(1):181-183. doi: 10.1016/j.tjog.2022.04.012. No abstract available. PMID 36720538
- [Result] Chen YY, Tsai CC, Lan KC, Ou YC. Preliminary report on the use of a levonorgestrel intrauterine system for the treatment of intermenstrual bleeding due to previous cesarean delivery scar defect. J Obstet Gynaecol Res. 2019 Oct;45(10):2015-2020. doi: 10.1111/jog.14060. Epub 2019 Aug 5. PMID 31381242
- [Result] Zhang J, Zhu C, Yan L, Wang Y, Zhu Q, He C, He X, Ji S, Tian Y, Xie L, Liang Y, Xia W, Mol BW, Huirne JAF. Comparing levonorgestrel intrauterine system with hysteroscopic niche resection in women with postmenstrual spotting related to a niche in the uterine cesarean scar: a randomized, open-label, controlled trial. Am J Obstet Gynecol. 2023 Jun;228(6):712.e1-712.e16. doi: 10.1016/j.ajog.2023.03.020. Epub 2023 Mar 17. PMID 36935068
- [Result] Zhang X, Yang M, Wang Q, Chen J, Ding J, Hua K. Prospective evaluation of five methods used to treat cesarean scar defects. Int J Gynaecol Obstet. 2016 Sep;134(3):336-9. doi: 10.1016/j.ijgo.2016.04.011. Epub 2016 Jun 30. PMID 27473332
- [Result] Zheng F, Chen S, Yang W, Li J, Huang Q, Qin H, Wei J, Lin J. Comparison of the efficacy of oral contraceptives and levonorgestrel intrauterine system in intermenstrual bleeding caused by uterine niche. Ginekol Pol. 2024;95(8):621-626. doi: 10.5603/GP.a2023.0067. Epub 2023 Jul 7. PMID 37417378